CLINICAL TRIAL: NCT05448508
Title: The Effects of Manual and Automatic Lancets on Pain and Stress in Newborn Capillary Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Meral Güven (Unknown); MSc Reyhan YALÇIN (Unknown); PhD Adem ASLAN (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Director, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TKP-2022-10664
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Newborn; Pain; Stress
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Lancet (Experimental): Manual lancet, needle tips and automatic lancets are used in the heel blood collection process. It has been reported that there may be complications arising from health professionals in the use of manual lancet or needle tip. In this study, an automatic lancet penetrating 2.4 mm-3 mm depth was used for safe puncture in term newborns.
  Interventions: Device: Automatic lancet
- Control (No Intervention): No intervention, routine maintenance performed

INTERVENTIONS:
Device: Automatic lancet — An automatic lancet, which can reach a depth of 2.4 mm-3 mm, was used for safe piercing in babies.
  Arms: Automatic Lancet

SUMMARY:
Heel blood sampling is a routine but painful procedure for newborns. A limited number of international studies have shown that automatic lancets are more effective with less pain and tissue damage than manual lancets.

In line with this information, this study was planned to investigate the effects of manual and automatic lancets on pain and stress in newborn capillary heel blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Postnatal age zero day
* Term newborn
* No congenital anomalies
* No advanced medical intervention at birth
* Infants not receiving oxygen or respiratory support

Exclusion Criteria:

* Legal guardian not giving consent to research

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The neo pain assessment scale | 12 week
  The neo scale was developed (2014) to assess pain and stress in premature and mature neonates. The Neo is a five-item scale including facial expression, breathing pattern, tone of extremities, hand and foot activity, and level of activity. The lowest and the highest scores obtainable from the scale are 0 and 10, respectively. As the score increases, stress and pain increase.
Crying time in second | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- AtaturkU, Yakutiye, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Kadiroglu T, Guven M, Yalcin R, Aslan A. The effects of manual and automatic lancet use on pain, stress, physiological parameters and crying duration during capillary heel blood collection in term neonates: a randomized controlled trial. BMC Nurs. 2025 Nov 18;24(1):1409. doi: 10.1186/s12912-025-04056-y. PMID 41254729